CLINICAL TRIAL: NCT04435522
Title: Open-Label Study of Maraviroc in Hospitalized Individuals Diagnosed With SARS-CoV-2
Brief Title: Maraviroc in Patients With Moderate and Severe COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1611471-1
Record Dates: First submitted 2020-06-15; First posted 2020-06-17 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2020-06

CONDITIONS: COVID
Keywords: Maraviroc; CCR5 Antagonist
MeSH Terms: interventions — Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Maraviroc Treatment (Experimental): Maraviroc 300 mg Twice Daily
  Interventions: Drug: Maraviroc

INTERVENTIONS:
Drug: Maraviroc — Maraviroc will be administered for seven days. Biomarkers of disease will be checked at time of enrollment, during and at the conclusion of therapy. The cytokine panel will consist of CCL5, IL-6, and Chitinase 3-like 1(Chi3l1).

SUMMARY:
Maraviroc, a C-C Chemokine Receptor 5 (CCR5) antagonist, is well-tolerated without significant side effects in its current use in patients with HIV. CCR5 antagonism prior to the 'second wave' of inflammatory mediator expression in SARS-CoV-2 may reverse lymphoid depletion and may alter cell trafficking of inflammatory cells, both increasing viral control capacity and dampening damage to lung tissue, respectively. This study seeks to establish whether one week of treatment with Maraviroc, used at its approved dosage for HIV, is safe and tolerable in patients with SARS-CoV-2.

DETAILED DESCRIPTION:
This pilot study seeks to establish that selective blockade of the CCR5/CCL5 axis as well as the potential anti-viral properties of Maraviroc may reduce disease severity. This proof-of-concept effort seeks to correlate differences in clinical outcomes to differential cytokine expression in the setting of CCR5 antagonism in patients infected with SARS-CoV-2. Maraviroc is FDA-approved for the treatment of CCR5-tropic HIV-1 and has a well-documented safety and tolerability record in previous trials in immunocompromised HIV patients. Maraviroc was not shown to have significant effect on the QT segment, can be delivered via oral formulation, and can be delivered safely to both patients with end-stage renal disease and dependence on hemodialysis12. For these reasons, Maraviroc is an ideal candidate to study as a potential therapy for hospitalized patients with moderate-to-severe COVID-19.

The primary objective is to establish whether Maraviroc, used at its approved dosage for HIV, is safe, tolerable, and effective in hospitalized patients with SARS-CoV-2. The secondary objective is to investigate the relationship between reduction of inflammatory markers (such as IL-6, CCL5, etc.) and clinical outcomes, including avoidance of respiratory decompensation and death.

This is a single-center, single-arm, open-label trial. Sixteen hospitalized patients will be enrolled. Screening data will be reviewed to determine subject eligibility. Subjects who meet all inclusion criteria and none of the exclusion criteria will be approached for consent prior to entering the study. Each subject will receive 7 days of Maraviroc twice daily. Each subject will have blood samples checked at time of enrollment (Day 0), Day 3, Day 7, and Day 15 or time of live discharge (whichever comes first) of the study. The total duration of subject participation will be five weeks. The total duration of the study is expected to be 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age at time of screening
* Documentation of a SARS-CoV-2 diagnosis as evidenced by positive SARS-CoV-2 PCR within twelve days at time of screening
* Chest radiography consistent with multi-focal pneumonia or air-space disease
* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.
* Subject able to safely swallow pills or receive Maraviroc through a nasogastric or orogastric tube.

Exclusion Criteria:

* Subjects who are pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Subjects with the presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data. This includes, but is not limited to, recent myocardial infarction in past 6 months, neurological, psychiatric, endocrine, or neoplastic diseases that are judged to interfere with participation in the study.
* Subjects with known diagnosis of human immunodeficiency virus infection (HIV)
* Subjects enrolled in another clinical trial (including one for COVID-19) that excludes participation in other trials or includes a potent CYP3A inhibitor or inducer (e.g. lopinavir-ritonavir).
* Subjects with ESRD or severe renal failure who are taking potent (moderate or strong) CYP3A inhibitors or inducers

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip A Chan, MD, Principal Investigator — Warren Alpert Medical School and School of Public Health, Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc Treatment: Maraviroc 300 mg Twice Daily
  Maraviroc: Maraviroc will be administered for seven days. Biomarkers of disease will be checked at time of enrollment, during and at the conclusion of therapy.
Period: Overall Study
Arm/Group | Maraviroc Treatment
Started | 9
Completed | 7
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Maraviroc Treatment
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Rate of Completion
Description: Rate of subjects who complete the 7-day course of Maraviroc (or shorter if discharged from hospital prior to 7 days) without discontinuation for serious adverse event or death.
Time Frame: 7 days
Population: Patients who received at least one dose of Maraviroc
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc Treatment
Number analyzed (Participants) | 7
Participants | 7

2. Primary Outcome: Clinical Improvement at Day 7
Description: Percent of patients at Day 7 from enrollment achieving reduction of two points on a seven-category ordinal scale (defined below).
  Ordinal scale: 1, not hospitalized with resumption of normal activities; 2, not hospitalized, but unable to resume normal activities OR hospitalized pending disposition, not requiring COVID-related care; 3, hospitalized, not requiring supplemental oxygen; 4, hospitalized, requiring supplemental oxygen; 5, hospitalized, requiring nasal high-flow oxygen therapy, noninvasive mechanical ventilation, or both; 6, hospitalized, requiring ECMO, invasive mechanical ventilation, or both; and, 7, death.
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Groups:
- Maraviroc Group: Single-arm group receiving Maraviroc for 7 days.
Arm/Group | Maraviroc Group
Number analyzed (Participants) | 7
Participants | 3

3. Secondary Outcome: Mortality
Description: 7-, 14- and 28-day all-cause-mortality
Time Frame: 28 days
Population: Population that received at least 1 dose of Maraviroc
Measure: Count of Participants; unit: Participants
Arm/Group | Maraviroc Treatment
Number analyzed (Participants) | 7
Participants
  7-Day Mortality | 0
  14-Day Mortality | 0
  28-Day Mortality | 0

4. Secondary Outcome: Median Time to >= 2 Point Improvement in Clinical Score.
Description: If no clinical improvement of >=2 points met by day 28, patient outcome censored
Time Frame: 28 Days
Measure: Median (Full Range); unit: Days
Arm/Group | Maraviroc Treatment
Number analyzed (Participants) | 7
Days | 8 [5 to 28]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 35 days from day of enrollement.
Arm/Group | Maraviroc Group
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 1/9
Other Adverse Events (participants affected / at risk) | 1/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc Group (N=9)
Death (Cardiac disorders) | 1 (1) — Subject death after withdrawl from study. Subject never received investigational agent.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maraviroc Group (N=9)
Nausea (Gastrointestinal disorders) | 1 (1)
Transaminitis (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-06): https://cdn.clinicaltrials.gov/large-docs/22/NCT04435522/Prot_SAP_000.pdf